CLINICAL TRIAL: NCT04463316
Title: GROWing Up With Rare GENEtic Syndromes ….When Children With Complex Genetic Syndromes Reach Adult Age
Brief Title: GROWing Up With Rare GENEtic Syndromes
Acronym: GROW UR GENES
Status: Recruiting | Type: Observational
Sponsor: dr. Laura C. G. de Graaff-Herder (Other)
Responsible Party: Sponsor-Investigator, dr. Laura C. G. de Graaff-Herder, Principal investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2018-1389
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Prader-Willi Syndrome; PWS-like Syndrome; Silver Russel Syndrome; Congenital Hypopituitarism; Klinefelter (XXY-)Syndrome; Congenital Adrenal Hyperplasia; XXXXY Syndrome; XXYY Syndrome; XXXX Syndrome (Tetra-X Syndrome); Disorders of Sex Development; Turner Syndrome; 46, XY DSD; Tuberous Sclerosis; Neurofibromatosis; Albright Hereditaire Osteodystrofie; Cornelia de Lange Syndrome; Saethre-Chotzen Syndrome; 17p- Deletiesyndrome; VCF Syndrome; POLR3A Mutatie; Ohdo Syndrome; Jacobsen Syndrome / 11 q Syndrome; Myrhe Syndrome; CHARGE Syndrome; 1q25-32 Deletie; Bardet Biedl Syndrome; Rett Syndrome; 22q11 Deletion Syndrome; Allan-Herndon-Dudley Syndrome; Kallmann Syndrome; Rare Bone Disorders; Noonan Syndrome; Williams-Beuren Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Klinefelter Syndrome; Adrenal Hyperplasia, Congenital; Tetrasomy X; Disorders of Sex Development; Turner Syndrome; Disorder of Sex Development, 46,XY; Tuberous Sclerosis; Neurofibromatoses; De Lange Syndrome; Acrocephalosyndactylia; DiGeorge Syndrome; Blepharophimosis syndrome Ohdo type; Jacobsen Distal 11q Deletion Syndrome; CHARGE Syndrome; Bardet-Biedl Syndrome; Rett Syndrome; 22q11 Deletion Syndrome; Allan-Herndon-Dudley syndrome; Kallmann Syndrome; Noonan Syndrome; Williams Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Retrospective file studies — No intevention, retrospective file study: medical history, laboratory values, additional tests, physical and psychological complaints.

SUMMARY:
Introduction Rare complex syndromes Patients with complex genetic syndromes, by definition, have combined medical problems affecting multiple organ systems, and intellectual disability is often part of the syndrome. During childhood, patients with rare genetic syndromes receive multidisciplinary and specialized medical care; they usually receive medical care from 3-4 medical specialists.

Increased life expectancy Although many genetic syndromes used to cause premature death, improvement of medical care has improved life expectancy. More and more patients are now reaching adult age, and the complexity of the syndrome persists into adulthood. However, until recently, multidisciplinary care was not available for adults with rare genetic syndromes. Ideally, active and well-coordinated health management is provided to prevent, detect, and treat comorbidities that are part of the syndrome. However, after transition from pediatric to adult medical care, patients and their parents often report fragmented poor quality care instead of adequate and integrated health management. Therefore, pediatricians express the urgent need for adequate, multidisciplinary adult follow up of their pediatric patients with rare genetic syndromes.

Medical guidelines for adults not exist and the literature on health problems in these adults is scarce. Although there is a clear explanation for the absence of adult guidelines (i.e. the fact that in the past patients with rare genetic syndromes often died before reaching adult age), there is an urgent need for an overview of medical issues at adult age, for 'best practice' and, if possible, for medical guidelines.

The aim of this study is to get an overview of medical needs of adults with rare genetic syndromes, including:

1. comorbidities
2. medical and their impact on quality of life
3. medication use
4. the need for adaption of medication dose according to each syndrome

Methods and Results This is a retrospective file study. Analysis will be performed using SPSS version 23 and R version 3.6.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rare syndromes or rare congenital diseases visiting the multidisciplinary outpatient clinic for patients with rare diseases at the department of endocrinology, internal medicine, Erasmus Medical Center.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex genetic syndromes
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence of physical health problems | 1 year
  For example: presence of hypertension, diabetes mellitus, hypercholesterolemia, scoliosis, sleep apnea, hypothyroidism, obesity, psychosis etc.
Laboratory values | 1 year
  For example: glucose, hemoglobin, hematocrit, thyroid hormone, TSH, estrogen, testosterone, LH, FSH, LDL-cholesterol, triglycerides, ASAT, ALAT, gamma-GT, etc
Physical and psychological complaints | 1 year
  For example: daytime sleepiness, obstipation, back pain, headache, behavioral problems, fatigue, nycturia, blurry vision, depressive symptoms, etc.
Medication use | 1 year
  Use of all medication

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon reasonable request.